CLINICAL TRIAL: NCT07142317
Title: The Impact of Plant Sterols on the Dietary Cholesterol-Induced Expression of GPR146: A Randomized Double-Blind Cross-Over Study
Brief Title: GPR146 and Cholesterol Metabolism
Acronym: GPR146
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 25-027
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: GPR146; Cholesin; Cholesterol metabolism; Gene expression; Postprandial study; Intestinal cholesterol absorption; Hepatic cholesterol synthesis; Plant sterols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cholesterol-poor, plant sterol-poor shake (Active Comparator): Participants will be given a mixed meal in the form of a cholesterol-poor, plant-sterol-poor shake.
  Interventions: Dietary Supplement: Cholesterol-poor, plant sterol-poor shake
- Cholesterol-rich, plant sterol-poor shake (Active Comparator): Participants will be given a mixed meal in the form of a cholesterol-rich, plant-sterol-poor shake.
  Interventions: Dietary Supplement: Cholesterol-rich, plant sterol-poor shake
- Cholesterol-rich plant sterol-rich shake (Experimental): Participants will be given a mixed meal in the form of a cholesterol-rich, plant-sterol-rich shake.
  Interventions: Dietary Supplement: Cholesterol-rich, plant sterol-rich shake

INTERVENTIONS:
Dietary Supplement: Cholesterol-poor, plant sterol-poor shake — The first arm is the cholesterol-poor arm, where participants will be given a mixed meal in the form of a cholesterol-poor, plant-sterol-poor shake which provides the lowest cholesterol absorption rate.
  Arms: Cholesterol-poor, plant sterol-poor shake
Dietary Supplement: Cholesterol-rich, plant sterol-poor shake — The second arm is the high-cholesterol arm, where participants will be given a mixed meal in the form of a cholesterol-rich, plant-sterol-poor shake, which provides the highest cholesterol absorption rate.
  Arms: Cholesterol-rich, plant sterol-poor shake
Dietary Supplement: Cholesterol-rich, plant sterol-rich shake — The third arm is the moderate-cholesterol arm, where participants will be given a mixed meal in the form of a cholesterol-rich, plant-sterol-rich shake, which provides the moderate cholesterol absorption rate.
  Arms: Cholesterol-rich plant sterol-rich shake

SUMMARY:
Blood cholesterol balance is regulated by an interplay between the small intestine and the liver. Recently, a new protein (cholesin) was discovered, which is secreted by intestinal cells after dietary cholesterol intake. Cholesin travels to the liver and binds to the GPR146 receptor. This inhibits cholesterol production in the liver. Because plant sterols lower blood cholesterol levels by reducing cholesterol absorption in the intestine, the investigators would like to understand the effects of plant sterols on GPR146. The investigator hypothesis is that the production of the GPR146 gene differs after adding plant sterols to a high-cholesterol diet compared to eating a high-cholesterol and low-cholesterol diet. The main objective of this study is to investigate whether the expression of the GPR146 gene in the blood of adults differs between three meals with different levels of cholesterol intake. The secondary objective of the study is to examine changes in the expression of cholesin, the LDL receptor (LDLR), and 3-hydroxy-3-methylglutaryl-CoA reductase (HMGCR) genes in the blood after these meals. Furthermore, changes in the expression of these genes, all of which play an important role in cholesterol metabolism, will be examined in intestinal cells.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged between 18-70 years
* BMI between 18.5-25.0 kg/m2
* Fasting serum total cholesterol (TC) <8.0 mmol/L and fasting serum triacylglycerol (TAG) <3 mmol/L
* Fasting plasma glucose (FBG) <7 mmol/L
* Systolic blood pressure <160 mmHg and diastolic blood pressure <100 mmHg
* Stable body weight (weight gain or loss of <3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study, and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Allergy or intolerance to any of the components of the study meal
* Familial hypercholesterolemia
* History of gastrointestinal surgery, including bariatric procedures such as sleeve gastrectomy, gastric bypass, gastric band, gastric balloon, or other major gastrointestinal surgeries that may affect digestion or absorption
* Current smokers
* Diabetic patients
* Pregnant and breastfeeding women
* Abuse of drugs
* More than 10 alcoholic consumptions per week for women and 14 for men
* Not willing to stop the use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigator for at least 1 week before the start of the study
* Use of medications to treat or affect blood pressure, lipid, or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1 month
* Severe medical conditions that might interfere with the study, such as: epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, autoinflammatory diseases, and rheumatoid arthritis
* Active cardiovascular disease, such as congestive heart failure, or a cardiovascular event, such as an acute myocardial infarction or a cerebrovascular accident

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The postprandial changes in GPR146 gene expression in peripheral blood mononuclear cells (PBMCs) after three dietary conditions. | At baseline (fasting; before the meal) and at 360 minutes (6-hours) postprandial
  The gene expression levels will be determined by messenger RNA (mRNA) quantification using the real-time reverse transcription polymerase chain reaction (RT-qPCR) method in PBMCs and reported as fold change (increase or decrease) relative to baseline.

SECONDARY OUTCOMES:
The postprandial changes in C7orf50, HMGCR, and LDLR gene expressions in peripheral blood mononuclear cells (PBMCs) after three dietary conditions. | At baseline (fasting; before the meal) and at 360 minutes (6-hours) postprandial
  The gene expression levels will be determined by messenger RNA (mRNA) quantification using the real-time reverse transcription polymerase chain reaction (RT-qPCR) method in PBMCs and reported as fold change (increase or decrease) relative to baseline
The postprandial changes in GPR146 and LDLR protein expressions in peripheral blood mononuclear cells after three dietary conditions. | At baseline (fasting; before the meal) and at 360 minutes (6-hours) postprandial
  The protein expression levels will be measured by fluorescence-activated cell sorting (FACS) analysis and reported as percentage of marker-positive cells and/or fold change in mean fluorescence intensity from baseline.

OTHER OUTCOMES:
The changes in small intestinal mucosal cells gene expression profiles of GPR146, C7orf50, HMGCR, and LDLR genes after the three meals | 6-hours postprandial
  The gene expression levels will be determined by messenger RNA (mRNA) quantification using the real-time reverse transcription polymerase chain reaction (RT-qPCR) method in small intestinal biopsy samples.
The postprandial response of serum triacylglycerol (TAG) and apolipoprotein B-48 (apoB-48) to the three meals | At intervals of 7 time-points during the postprandial period (0-6 hours)
  Serum TAG will be measured spectrophotometrically, and apoB-48 will be quantified by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Due to data protection and participants' confidentiality, this will be decided by the principal investigator based on a reasonable request.